CLINICAL TRIAL: NCT03876145
Title: A Comparison of Four Methods of Ovarian Stimulation With GnRH Antagonist in Patients With Polycystic Ovarian Syndrome in Royan Institute; A Randomized Controlled Clinical Trial
Brief Title: The Four Methods of Ovarian Stimulation in Patients With Polycystic Ovarian Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Female Infertility
Record Dates: First submitted 2019-02-25; First posted 2019-03-15 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2019-02

CONDITIONS: Polycystic Ovary Syndrome; Ovarian Hyperstimulation Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Ovarian Hyperstimulation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Minimal ovarian stimulation with rec-FSH (Experimental): The group of minimal ovarian stimulation that will receive 100 mg clomiphene citrate every day from Day 3 to Day 7 of the menstrual cycle and then will be treated with 150 International Unit (IU) Gonal-f (Follitropin alfa, Merck Serono, Germany) after the seventh day.
  Interventions: Other: Minimal ovarian stimulation
- Minimal ovarian stimulation with HMG (Experimental): The group of minimal ovarian stimulation that will receive 100 mg clomiphene citrate every day from Day 3 to Day 7 of the menstrual cycle and then will be treated with 150 IU Merional (Highly Purified Menotropin، IBSA، Switzerland) after the seventh day.
  Interventions: Other: Minimal ovarian stimulation
- Mild ovarian stimulation with rec-FSH (No Intervention): The group of mild ovarian stimulation that will receive 150 IU Gonal-f (Follitropin alfa, Merck Serono, Germany) daily from Day 3 of the menstrual cycle.
- Mild ovarian stimulation with HMG (No Intervention): The group of mild ovarian stimulation that will receive 150 IU Merional (Highly Purified Menotropin، IBSA، Switzerland) daily from Day 3 of the menstrual cycle.

INTERVENTIONS:
Other: Minimal ovarian stimulation — After obtaining informed consent to participate in the study, the subjects will be randomly divided into the following 4 groups: The group of minimal ovarian stimulation with rec-FSH or HMG. The group of mild ovarian stimulation with rec-FSH or HMG. In all 4 experimental groups, after reaching at least three follicles the size of 12 millimeters (mm), daily administration of 0.25 milligram (mg) Cetrotide (antagonist GnRH) will be started and after reaching at least three follicles the size of 17 mm, 500 microgram Ovitrelle (recombinant Human curionic gonadotropin) will be prescribed. 36 hours later, ovulation process will be done. On the day of Ovitrelle administration, serum levels of estradiol and progesterone will be also evaluated. Based on the patient's condition and the quality of obtained oocytes and embryos, 2 embryos will be transferred.
  Arms: Minimal ovarian stimulation with HMG; Minimal ovarian stimulation with rec-FSH

SUMMARY:
This study is a randomized controlled clinical trial to compare the pregnancy outcomes of mild and minimal stimulation in infertile women with polycystic ovarian syndrome. The study population consisted of all infertile women with polycystic ovary syndrome based on Rotterdam criteria who have not succeed to achieve fertility despite multiple treatments such as drug therapy, laparoscopic surgery, and the frequent failure of induction therapy using gonadotropins and are now candidate for in vitro fertilization (IVF) or intra cytoplasmic sperm injection (ICSI) in Reproductive Biomedicine Research Center, Royan institute, Tehran Iran.

DETAILED DESCRIPTION:
An overview of the history of assisted reproductive technologies such as IVF and ICSI that are based on the process of ovulation stimulation, suggests that although this process was initially welcomed with the aim of achieving a large number of oocytes and embryos, consequences such as low quality of obtained oocytes and embryos, failure in achieving the desired results in fertility of treated patients, and the incidence of adverse effects such as ovarian hyper stimulation syndrome have made researchers re-examine the process of ovulation stimulation. Hence, mild ovulation stimulation method has been introduced to the field of assisted reproductive techniques (ART) in recent years. This method includes the prescription of low doses of gonadotropins or shorter duration of its administration in the ovulation stimulation cycle. Mild ovulation method has advantages such as reduction of the physical, mental, and financial risks of treatment which can improve the quality assisted reproductive services provided for infertile couples.

Several studies have confirmed the efficiency of this method of ovulation stimulation as a way for improving the quality of the ovulation process and achieving desirable results in fertility. However, the important and interesting point in studies conducted in this area, particularly on IVF and ICSI cycles, is that the application of this method has been mostly investigated in normal populations and, after the approval of its efficiency, it has been recommended to be used in patients with poor or high ovarian response. It should be also mentioned that efficiency of this method in patients with poor ovarian response has been evaluated in a few studies, while in patients with high ovarian response such as those suffering from polycystic ovary syndrome, only few studies have been conducted in patients with a history of ovarian hyper stimulation syndrome. On the other hand, in many cases, the efficiency of mild ovulation stimulation, in which lower doses or shorter durations of gonadotropin administration are desired, has been investigated, and the application of minimal ovulation stimulation method, in which the use of clomiphene citrate is also included besides lower doses or shorter durations of gonadotropin administration, has been studied in a few cases.

In addition to the dose and duration of gonadotropin administration, another important point in achieving the desired results of treatment using the ovulation stimulation cycles is the type of gonadotropin. The studies conducted on the comparison of recombinant-FSH (rec-FSH) and Human Menopausal Gonadotropin (HMG) types of gonadotropin indicate the superiority of HMG gonadotropins, as the results show that the administration of HMG gonadotropins will lead to achieving fewer but high quality oocytes and embryos. By contrast, rec-FSH application puts the patients at increased risk of ovarian hyper stimulation syndrome. However, the interesting and important point in most of these studies is that this comparison has been drawn in long-term treatment cycles, while few studies have been conducted on antagonist treatment cycles which do not fully corroborate the results obtained from long-term cycles.

According to what mentioned above, the present research aims to study the efficiency of minimal ovulation stimulation method in the treatment of infertile patients with poly cystic ovarian syndrome (PCOS) and also the effect of gonadotropin type on treatment cycles with antagonist gonadotropin-releasing hormone (GnRH). It is hoped that the findings of the present research provide solutions for improving the quality of infertility treatment in PCOS patients, who currently undergo IVF or ICSI as a last resort.

ELIGIBILITY:
Inclusion Criteria:

1. Infertile women with polycystic ovary syndrome based on Rotterdam criterion
2. 20<Age<38
3. BMI<30
4. Non recurrent miscarriage
5. Non endocrine, hematologic and autoimmune disorders
6. Non chromosomal and genetic abnormalities
7. Non uterine anomalies, surgical history, endometriosis, adenomyosis, hydrosalpinx, uterine fibroids
8. Non azoospermia

Exclusion Criteria:

1. Patient's tendency for withdrawal

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-11-12 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Fertilization rate | 16-18 hours after start of IVF or ICSI, which occurs on day of oocyte pick-up (34-36 hours after hCG administration [approximately Stimulation Day 10]).
  The ratio of 2 pronuclear to total number of injected oocytes.
Implantation rate | 4 weeks after embryo transfer
  The ratio of total number of observed gestational sacs to total number of transferred embryos.
Clinical pregnancy rate | 4 weeks after embryo transfer
  The observation of gestational sac with heart beat by using trans-vaginal ultrasound.

SECONDARY OUTCOMES:
ovarian hyper stimulation syndrome (OHSS) rate | Up to approximately 2 month after oocyte pick-up (34-36 hours after hCG administration [approximately Stimulation Day 10]).
  Total number of cases with symptoms of ovarian hyper-stimulation syndrome.
Total number of retrieved oocytes | Day of oocyte pick-up, 34-36 hours after human curionic gonadotropin (hCG) administration (approximately Stimulation Day 10).
  Total number of obtained oocytes which reported by embryologist.
Quality of retrieved oocytes | Day of oocyte pick-up, 34-36 hours after hCG administration (approximately Stimulation Day 10).
  Total number of Meta-phase II oocytes which reported by embryologist.

CONTACTS AND LOCATIONS:
Overall Officials: Firoozeh Ghaffari, M.D., Study Director — Department of Endocrinology and Female Infertility, ACECR, Tehran, Iran.; Azar Yahyaei, M.Sc., Principal Investigator — Department of Endocrinology and Female Infertility, ACECR, Tehran, Iran.
Locations (1):
- Royan Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yahyaei A, Vesali S, Ghaffari F. Introduce an optimal method of ovarian stimulation in the polycystic ovarian syndrome affected: a randomized controlled trial. BMC Womens Health. 2023 Jun 20;23(1):323. doi: 10.1186/s12905-023-02473-2. PMID 37340371